CLINICAL TRIAL: NCT00485004
Title: FOcal Type In-stent Restenosis After Drug-Eluting Stent Implantation Treated by CUtting Balloon Angioplasty Versus Sirolimus-Eluting Stent
Brief Title: Focal In-stent Restenosis After Drug-Eluting Stent
Acronym: FOCUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070041
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: In Stent Restenosis
Keywords: Coronary artery disease; Stent; Angioplasty
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cutting balloon (Experimental): Cutting balloon
  Interventions: Device: Cutting balloon; Device: Sirolimus-eluting stent
- Sirolimus-eluting stent (Active Comparator): Sirolimus-eluting stent
  Interventions: Device: Cutting balloon; Device: Sirolimus-eluting stent

INTERVENTIONS:
Device: Cutting balloon — Cutting balloon
Device: Sirolimus-eluting stent — Sirolimus-eluting stent

SUMMARY:
To evaluate the optimal management of focal in-stent restenosis after drug-eluting stent implantation with sirolimus-eluting implantation versus cutting balloon angioplasty

DETAILED DESCRIPTION:
Following angiography, patients with focal DES restenosis (lesion length ≤ 10mm) with diameter stenosis >50% by visual estimation have documented myocardial ischemia or symptoms of angina, and eligible for PCI without any exclusion criteria will be randomized 1:1 to: a) Cypher stent vs. b) Cutting balloon angioplasty. All patients will be followed for 1 year. Angiographic follow-up at 9-months is mandatory.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age.
2. Restenosis after drug-eluting stents (>50% by visual estimate)
3. Lesion length < 10 mm (focal ISR)
4. Patients with stable (CCS class 1 to 4) or acute coronary syndromes (unstable angina pectoris Braunwald class IB, IC, IIB, IIC, IIIB, IIIC or NSTEMI) or patients with atypical chest pain or without symptoms but having documented myocardial ischemia, amenable to stent-assisted percutaneous coronary intervention
5. The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications:

   * Heparin
   * Aspirin
   * Both Clopidogrel and TIclopidine
   * Sirolimus eluting stent
   * Stainless steel and/or
   * Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled).
2. Systemic (intravenous) Sirolimus use within 12 months.
3. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
4. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
5. Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
6. Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL.
7. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
8. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
9. Patients with EF<30%.
10. Acute MI patients within symptom onset < 12 hours needing primary angioplasty
11. Creatinine level 3.0mg/dL or dependence on dialysis.
12. Severe hepatic dysfunction (AST and ALT 3 times upper normal reference values).
13. Patients with left main stem stenosis and left main in-stent restenosis created by DES(>50% by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Binary In-segment Restenosis | At 9 months angiographic follow-up

SECONDARY OUTCOMES:
Composite end-point of death, myocardial infarction, or target vessel revascularization | At 9-month after index procedure
Stent thrombosis | In-hospital, 30 days, 9 months, and 1year
Late luminal loss | at 8 month angiographic follow-up
Procedural success defined as achievement of a final diameter stenosis of <30% by QCA using any percutaneous method, without the occurrence of death, Q wave MI, or repeat revascularization of the target lesion | during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (15):
- South Korea (15):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Choeng Ju St.Mary's Hospital, Choeng Ju
  - Kangwon National University Hospital, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Gangneung
  - DongGuk University Gyongju Hospital, Gyongju
  - Chonbuk National University Hospital, Jeonju
  - Kwangju Christian Hospital, Kwangju
  - Inje University Pusan Paik Hospital, Pusan
  - Hallym University Sacred Heart Hospital,, Pyeongchon
  - Asan Medical Center, Seoul
  - Hangang Sacred Heart Hospital, Seoul
  - Kyungsang University Hospital, Seoul
  - Seoul Veterans Hospital, Seoul
  - Ulsan University Hospital, Ulsan